CLINICAL TRIAL: NCT01250743
Title: An Open-Label Pilot Study of the Safety, Tolerability and Anti-Viral Activity of High Dose Intravenous Ascorbic Acid in Patients Chronically Infected With Hepatitis C Virus Genotype 1, Who Have Failed Prior Therapy With Interferon-alpha and Ribavirin
Brief Title: A Pilot Study of High-Dose, Intravenous Ascorbic Acid (Vitamin C) to Treat Hepatitis C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Health Innovations, Frontier Research Institute (Other)
Responsible Party: Michael A Catalano MD, Research Director, Health Innovations, Frontier Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRI-101
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2010-11

CONDITIONS: Hepatitis C
Keywords: genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ascorbic Acid (Vitamin C) (Experimental)
  Interventions: Dietary Supplement: ascorbic acid (vitamin C)

INTERVENTIONS:
Dietary Supplement: ascorbic acid (vitamin C) — intravenous vitamin C, 25 to 100 grams, once or twice a week, for five months
  Other Names: Vitamin C

SUMMARY:
The purpose of this pilot study is to learn whether high doses of ascorbic acid (vitamin c), given intravenously to patients with chronic hepatitis due to infection with the genotype 1 version of the hepatitis C virus, are safe, well-tolerated and able to reduce the amount of virus circulating in the patients' blood.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) chronically infects 1% to 3% of the world's population, including about 3.9 million infected patients in the United States, with an estimated 36,000 new cases in the US each year. 70-85% of infected individuals develop a chronic infection complicated by chronic liver disease during the next 20 to 30 years, which is the tenth leading cause of death in the US. HCV is implicated in the development of hepato-cellular carcinoma. Chronic HCV hepatitis is the most frequent reason for liver transplantation. HCV genotype 1 is the most common genetic variant of HCV causing HCV hepatitis in the US. It responds less well to conventional anti-HCV treatment than the other HCV genotypes, so that 60% of genotype 1 patients fail conventional therapy due to the virus's resistance to treatment and/or due to toxic side effects of the therapy.

Extracellular levels of ascorbic acid (vitamin c) attainable only by high-dose, intravenous administration, are reported to have in vitro and in vivo anti-cancer and anti-viral effects in humans and animals. Ascorbic acid briefly generates extracellular hydrogen peroxide, an oxidative stress specifically toxic to cancer cells and cells infected with viruses, including HCV, but not to normal cells. High-dose, intravenous ascorbic acid has been given to large numbers of patients, particularly cancer patients, with anecdotal reports of good safety and occasional benefit. Given the foregoing, the investigators propose that there is sufficient rationale for a careful pilot study of the safety and anti-viral efficacy of infused ascorbic acid in HCV genotype 1 hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* hepatitis C, genotype 1
* failed treatment with interferon-alpha and ribavirin
* abstain from alcohol consumption for the duration of the study

Exclusion Criteria:

* cirrhosis
* decompensated liver disease
* glucose6phosphate dehydrogenase deficiency
* AST or ALT more than 5 times upper limit of normal
* platelets less than 125,000
* diabetes mellitus
* alcohol and/or drug abuse within 1 year of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
number of participants with adverse events as a measure of safety and tolerability | 6 months
  clinical and/or laboratory adverse events

SECONDARY OUTCOMES:
anti-viral efficacy | 6 months
  measured by reduction of circulating hepatitis C viral levels
aspartate aminotransferase (AST or SGOT) | 6 months
  reduced circulating levels of AST (or SGOT), as a measure of liver inflammation
alanine aminotransferase (ALT or SGPT) | 6 months
  reduced circulating levels of ALT (or SGPT), as a measure of liver inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne A Drisko, MD, Principal Investigator — University of Kansas Medical Center; Michael A Catalano, MD, Study Director — Frontier Research Institute/Health Innovations; Terry A Grossman, MD, Study Chair — Frontier Research Institute/Health Innovations
Locations (1):
- University of Kansas Medical Center, Department of Integrative Medicine, Kansas City, Kansas, United States

REFERENCES:
- [Background] Choi J, Lee KJ, Zheng Y, Yamaga AK, Lai MM, Ou JH. Reactive oxygen species suppress hepatitis C virus RNA replication in human hepatoma cells. Hepatology. 2004 Jan;39(1):81-9. doi: 10.1002/hep.20001. PMID 14752826
- [Background] Chen Q, Espey MG, Krishna MC, Mitchell JB, Corpe CP, Buettner GR, Shacter E, Levine M. Pharmacologic ascorbic acid concentrations selectively kill cancer cells: action as a pro-drug to deliver hydrogen peroxide to tissues. Proc Natl Acad Sci U S A. 2005 Sep 20;102(38):13604-9. doi: 10.1073/pnas.0506390102. Epub 2005 Sep 12. PMID 16157892